CLINICAL TRIAL: NCT03146780
Title: Clinical Evaluation of Digital Versus Conventional Impressions Part I: Marginal and Internal Fit
Brief Title: Digital vs Conventional Impressions Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Konstantinos Chochlidakis, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RSRB#00065524
Record Dates: First submitted 2017-05-01; First posted 2017-05-10 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Dental Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conventional (Placebo Comparator)
  Interventions: Procedure: Conventional impression
- Digital 1 (Active Comparator)
  Interventions: Procedure: Digital Scan 1
- Digital 2 (Active Comparator)
  Interventions: Procedure: Digital Scan 2
- Digital 3 (Active Comparator)
  Interventions: Procedure: Digital Scan 3

INTERVENTIONS:
Procedure: Conventional impression — A dental impression is a negative imprint of hard (teeth) and soft tissues in the mouth from which a positive reproduction (or cast) can be form using alginate material. They are made by using a container which is designed to roughly fit over the dental arches ("trays").
  Arms: Conventional
Procedure: Digital Scan 1 — Direct intra-oral digital scans using Sirona Omnicam software.
  Arms: Digital 1
Procedure: Digital Scan 2 — Direct intra-oral digital scans using Planmeca Planscan software.
  Arms: Digital 2
Procedure: Digital Scan 3 — Direct intra-oral digital scans using 3M True Definition software.
  Arms: Digital 3

SUMMARY:
This study aims to compare how a single cap best fit on a tooth that is fabricated with digital and conventional impression techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age of patient ≥ 18 years old
* Good oral hygiene and compliance
* In need of a single full-coverage crown on any vital premolar or first molar tooth
* Opposing tooth is free of indirect restoration (crown)
* Asymptomatic tooth free of pathology
* No requirement for additional treatment (endodontic treatment, post and core, crown lengthening)
* Anticipated supragingival or equigingival crown margin
* Anticipated crown margin on natural tooth structure
* Adequate abutment height after tooth preparation (minimum 4mm)

Exclusion Criteria:

* Age of patient less than 18 years old
* Poor oral hygiene and calculus on sample teeth
* In need of a single full-coverage crown on tooth other than a vital premolar or first molar tooth
* Opposing tooth is restored with indirect restoration
* Periapical or periodontal pathology
* Anticipated pulp exposure or need for additional treatment (endodontic treatment, post and core, crown lengthening)
* Anticipated subgingival crown margin
* Anticipated crown margin on direct restoration
* Inadequate abutment height after tooth preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with a correctly fitted prosthesis | From impression stage to crown delivery, approximately four weeks. There are no follow up visits once crown is delivered.
  Correct fit assessed by clinical assessment of internal and marginal crown fit.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No